CLINICAL TRIAL: NCT04544683
Title: The Effectiveness of Cervical Transforaminal Epidural Steroid Injection for the Treatment of Cervical Radicular Pain: A Prospective Cohort Study.
Brief Title: Effectiveness of Cervical Transforaminal Epidural Steroid Injection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Zack McCormick, Zachary McCormick, MD FAAPMR, Associate Professor, Director of Clinical Spine Research, Director of Interventional Spine and Musculoskeletal Medicine Fellowship, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB 116040
Record Dates: First submitted 2020-08-28; First posted 2020-09-10 (Actual); Results first posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-03

CONDITIONS: Cervical Radiculopathy; Cervical Spondylosis; Disk, Herniated
Keywords: Transforaminal Epidural Injection
MeSH Terms: conditions — Radiculopathy; Spondylosis; Intervertebral Disc Displacement | interventions — dexamethasone 21-phosphate

STUDY DESIGN:
Intervention Model Description: Through a research questionnaire, pre-procedure and post procedure NRS pain score for both neck and arm we will obtain data regarding cervical epidural steroid injections via a transforaminal approach for research purposes only. Also current pain medications of patient throughout treatment will be obtained for research purposes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cervical Pain for 6 months or less and scheduled for TFESI (Other): Participants who meet inclusion and exclusion criteria will be enrolled into the study after consenting to and before receiving a first cervical TFESI. The baseline examination and all baseline questionnaires will be completed within 2 weeks before the first cervical TFESI. Participants will be given a daily pain diary chart to record NRS and percentage improvement during the 1st month post-injection. Participants will be contacted in the 1st week post-injection with a standardized questionnaire about their symptoms and a reminder about the 4 week (+/- 1 week) post-injection follow up. Routine scheduled follow-up by clinic visit or telephone call will occur at 4 weeks (+/- 1 week), 8 weeks (+/- 2 weeks), 3 months (+/- 2 weeks), 6 months (+/- 1 month), and 12 months (+/- 1 month), at which times all follow-up measures will be obtained.
  Interventions: Drug: Cervical Transforaminal Epidural Injection with dexamethasone sodium phosphate

INTERVENTIONS:
Drug: Cervical Transforaminal Epidural Injection with dexamethasone sodium phosphate — Transforaminal epidural steroid injection: Injection of 1 to 2 mL of 1% lidocaine to the skin and subcutaneous tissues, a 25-gauge spinal needle will be placed at the level and side of radicular pathology, based on clinical correlation of symptoms/signs and magnetic resonance imaging findings. Advancement to the appropriate target position in the neuroforamen will be performed under fluoroscopic guidance. Satisfactory target position achieved and confirmed in both anterior-posterior and oblique views, 0.5 to 1 mL of contrast will be injected under live fluoroscopic observation with or without digital subtraction angiography depending on suggestion of vascular uptake. Upon confirmation of a satisfactory epidural contrast pattern without vascular uptake, the injectate will be delivered: dexamethasone sodium phosphate 1mL (10mg/mL) and 0.5 ml of 1% preservative-free lidocaine (total volume 1.5 mL).

SUMMARY:
Study Purpose:

This study is intended to monitor outcomes for 1 year following cervical TFESI. Based on current clinic volume and enrollment rates into a current study of cervical epidural injections that is nearing completion, we conservatively estimate a study enrollment period of 18 months and a total period of 2.5 years from enrollment to final follow-up data collection. If the study were to theoretically start enrolling in July 2019, we would anticipate completion by February 2022.

Objectives:

1. Determine the proportion of patients with an 80% or greater improvement in arm and neck numerical rating scale pain (NRS) score following an initial cervical transforaminal steroid injection (TFESI) at 4 weeks post-injection and the duration of response up to 12 months.
2. Determine the proportion of patients with a 50%-79% improvement in arm and neck NRS score following an initial cervical TFESI at 4 weeks post-injection and the duration of response up to 12 months.
3. Determine the proportion of patients with less than 50% improvement in arm and neck NRS score following an initial cervical TFESI at 4 weeks post-injection and the duration of response up to 12 months.
4. Determine the proportion of patients with an initial injection plus up to 3 additional injections that maintain 80% or greater, as well as 50-79%, improvement in arm and neck NRS score for up to 12 months.
5. Determine the proportion of patients with a clinically significant change in function defined by a minimally clinically significant change (MCIC) (≥10 point improvement ) or 30% improvement in Neck Disability Index (NDI) score following an initial cervical TFESI at 4 weeks post-injection and the duration of response up to 12 months.
6. Determine the proportion of patients with clinically significant improvement in the Medication Quantification Scale (MQS III) score (≥6.8 point change , equivalent to 10 oral morphine equivalents ) following an initial cervical TFESI at 4 weeks post-injection and the duration of response up to 12 months.

6. Determine the proportion of patients with clinically significant improvement in the categorical EuroQol 5 Dimensions tool (EQ-5D) defined by ≥0.03 following an initial cervical TFESI at 4 weeks post-injection and the duration of response up to 12 months.

7. Compare patient demographic, clinical, and imaging characteristics between response groups and perform predictive modeling to better understand variables that increase the likelihood of a successful clinical outcome.

8. Report adverse effects.

DETAILED DESCRIPTION:
Background and Project Justification: Neck pain is now the fourth leading cause of years lost to disability, shortly after back pain, depression, and arthralgia. Cervical radiculopathy, a common cause of neck and radiating arm pain, is estimated to afflict 83:100,000 individuals yearly. Age-related cervical spondylosis and disc herniation are the most common causes, with the C6 and C7 nerve roots most frequently affected. In general, patients who experience new onset radicular pain tend to improve within 4-6 months, with complete recovery in over 80% of patients by 24-36 months. However, a significant proportion of patients experience severe pain and associated functional impairment despite conservative care, which often prompts physician directed interventions.

Cervical transforaminal epidural steroid injection (TFESI) is a target-specific treatment for refractory radicular pain. Analgesic mechanisms for epidural steroid administration include reducing inflammation at the nerve root, reducing nociceptive input from somatic nerves, stabilization of neural membranes, and blockade of C fiber activity in the dorsal root ganglion . Previously, this procedure was associated with rare but catastrophic neurologic injury, though to be related to inadvertent deposit of particulate steroid into the vertebral artery or radiculomedullary arteries, both of which traverse through or close to the cervical neuroforamina . Since the physician community has adopted new guidelines that include the use of only non-particulate steroid during cervical TFESI , neurologic infarction has not been reported in the literature. When the Spine Intervention Society (SIS) clinical practice guidelines are employed, large cohort study demonstrates zero prevalence of serious complications associated with this procedure .

While high-quality outcome literature demonstrates both efficacy and effectiveness for analogous use of this intervention in the lumbar spine, far fewer studies have addressed clinical outcomes associated with cervical TFESI in which appropriate procedure technique , outcome measurement, data analysis, and results interpretation have been reported . Outcome literature reporting on the use of cervical TFESI is limited by small sample size, retrospective design with loss of follow-up, lack of categorical data analysis, and a failure to stratify results by demographic and clinical variables that potentially influence pain and functional outcomes. Further, outcome literature reports on the effect of particulate steroid injectate during cervical TFESI is no longer relevant to appropriate clinical practice in the context of unequivocal guidelines. Pragmatic studies with a cervical TFESI arm in which dexamethasone was use do allow for some insight regarding success rates associated with this procedure; calculates of success rates in these studies arms demonstrate responder rates of 60% achieving >50% pain relief (CI95 35-85%) at 4 weeks, 55% achieving >50% (CI95 43-67%) at 8 weeks, and 65% achieving >50% at 12 weeks (CI95 48-81%). These responder rates are encouraging, but limited by wide 95% confidence intervals due to small sample size. Prior systematic review has concluded that the evidence for treatment benefit of radicular pain by cervical TFESI is of very low quality due to multiple limitations in study design introducing risk of bias, but does overall suggest approximately 50% patients experience 50% relief of radicular pain for at least 4 weeks after cervical TFESI.

Additional clinical outcome literature is needed, particularly given recent policy decisions, such as that of Oregon State in relation to ending coverage of epidural steroid injections at any spinal level. Without expansion of the evidence-basis for this important procedure, there is a risk that this treatment option may be taken away from patients suffering from cervical radicular pain by further policy change. A sham-controlled trial, similar to the Ghahreman study, would be ideal; however, due to cost considerations germane to a study designed and conducted in a manner that would prevent any possible criticism from the larger medical community, we instead propose a high-quality, large prospective cohort study as a significant contribution to the literature. Even the best designed trials, such as Dreyfuss' 2006 study, have been underpowered to definitively demonstrate effectiveness; notably, the lower bound of the 95% confidence interval of the proportion of treatment responders in this study was 35%. The investigators aim to conduct a large enough cohort study narrow the 95% confidence interval of the proportion of responders substantially. Preliminary data from our center demonstrates a responder rate of 55% at 4-week follow-up (n=22), based on a definition of ≥50% improvement in index pain (Appendix A). These data represent analysis of consecutive patients who underwent cervical TFESI for unilateral radicular pain as a part of a different prospective outcome study at our center, nearing completion. This responder rate represents a conservative estimate of what might be expected in the proposed work, as the current study includes less stringent inclusion and exclusion criteria.

Further, the investigators intend to use the results of this study as foundational data from which to propose a randomized controlled study through a large federal funding mechanism. It is imperative that such a trial be conducted by investigators who are experienced with this procedure and understand the appropriate standards for the design and interpretation of the results of a study of a treatment intervention for pain. Our spine research group is well-positioned for this, and we absolutely welcome the input and mentorship of the Spine Intervention Society Research Division, Board of Directors, and other leadership towards this mutual goal.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18-80 capable of understanding and providing consent in English and capable of complying with the outcome instruments used.
* Arm pain or shoulder girdle pain/periscapular pain with or without neck pain with duration less than or equal to 6 months.
* 3-day average numeric pain rating score (NRS) for arm pain or shoulder girdle/periscapular pain of at least 4/10 at baseline evaluation, with neck pain score not exceeding arm and/or shoulder girdle/periscapular pain score.
* MRI (or CT if MRI not available) shows either a one level cervical disc herniation, disc osteophyte complex or degenerative foraminal stenosis, corresponding in side and location with predominately unilateral radicular pain, with or without neurological deficits. MRI may show degenerative changes at other levels.
* Patient consents to treatment with epidural injection in a shared decision-making process with the treating physician.
* Pain duration of at least 6 weeks or more.

Exclusion Criteria:

* Those receiving remuneration for their pain treatment (e.g., disability, worker's compensation).
* Those involved in active litigation relevant to their pain.
* The patient is incarcerated.
* Neck pain is greater than arm pain or shoulder girdle/periscapular pain.
* Bilateral radicular signs/symptoms (< 90% laterality of pain intensity, or bilateral neurological signs).
* BMI>35.
* Prior epidural steroid injections for treatment of current episode.
* Those unable to read English and complete the assessment instruments.
* Spondylolisthesis at the involved or adjacent segments.
* Systemic inflammatory arthritis (e.g., rheumatoid, lupus).
* Addictive behavior, severe clinical depression, or psychotic features.
* Possible pregnancy or other reason that precludes the use of fluoroscopy.
* Treatment of infection with antibiotics within the past 7 days.
* Progressive motor deficit and/or clinical signs of myelopathy.
* History of prior cervical spine surgery.
* Medical conditions causing significant functional disability (e.g., stroke, COPD)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2023-12-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cervical Pain for 6 Months or Less and Scheduled for TFESI: Consenting participants who met eligibility criteria were enrolled into the study. The baseline examination and all baseline questionnaires were completed within 2 weeks before the first cervical TFESI. All follow-up measures were obtained at routine scheduled follow-up by clinic visit or telephone occurred at 1 month (+/- 1 week), 3 months (+/- 2 weeks), 6 months (+/- 1 month), and 12 months (+/- 1 month).
  Cervical Transforaminal Epidural Injection with dexamethasone sodium phosphate: Transforaminal epidural steroid injection: Injection of 1 to 2 mL of 1% lidocaine to the skin and subcutaneous tissues, a 25-gauge spinal needle will be placed at the level and side of radicular pathology, based on clinical correlation of symptoms/signs and magnetic resonance imaging findings. Advancement to the appropriate target position in the neuroforamen will be performed under fluoroscopic guidance. Satisfactory target position achieved and confirmed in both anterior-posterior and oblique views, 0.5 to 1 mL of contrast will be injected under live fluoroscopic observation with or without digital subtraction angiography depending on suggestion of vascular uptake. Upon confirmation of a satisfactory epidural contrast pattern without vascular uptake, the injectate will be delivered: dexamethasone sodium phosphate 1mL (10mg/mL) and 0.5 ml of 1% preservative-free lidocaine (total volume 1.5 mL).
Period: Overall Study
Arm/Group | Cervical Pain for 6 Months or Less and Scheduled for TFESI
Started | 33
1 Month Follow-up | 30
3 Month Follow-up | 29
6 Month Follow-up | 26
12 Month Follow-up | 25
Completed | 25 (Of the 33 enrolled participants, 25 completed the study. The 8 individuals who didn't complete the study were included in worst-case scenario analyses as treatment failures.)
Not Completed | 8
Not completed — Lost to Follow-up | 2
Not completed — Underwent cervical spine surgery | 6

BASELINE CHARACTERISTICS:
Arm/Group | Cervical Pain for 6 Months or Less and Scheduled for TFESI
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Duration of Pain [Count of Participants; unit: Participants]
  6 weeks to 3 months | 13
  >3 months up to 6 months | 20
Arm Pain Numeric Rating Scale [Mean (Standard Deviation); unit: units on a scale] — Arm pain was defined and explained to participants as being discomfort experienced in the periscapular, shoulder, upper arm, lower arm, or hand. Participants rated their arm pain intensity on an 11-point Numeric Rating Scale ranging from 0 to 10, with 0 representing "no pain at all" and 10 representing "the worst pain imaginable".
  units on a scale | 6.5 (1.4)
Neck Pain Numeric Rating Scale [Mean (Standard Deviation); unit: units on a scale] — Neck pain was defined as pain localized to the cervical spine. Participants rated their neck pain intensity on an 11-point Numeric Rating Scale ranging from 0 to 10, with 0 representing "no pain at all" and 10 representing "the worst pain imaginable".
  units on a scale | 4.5 (2.9)
Neck Disability Index (NDI-5) [Mean (Standard Deviation); unit: units on a scale] — The 5-Item Neck Disability Index (NDI-5) is an assessment tool measuring patients' self-reported functional limitations due to neck pain. The range of possible scores is 0 to 24, with higher scores indicating greater functional impairment in activities of daily living.
  units on a scale | 9.4 (3.9)
EuroQol Health-Related Quality of Life (EQ-5D) [Mean (Standard Deviation); unit: units on a scale] — The EuroQol Health-Related Quality of Life 5-Dimension (EQ-5D) is an instrument used in clinical and research settings to assess overall quality of life across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Scores are reported as an index ranging from 0 to 1, where 0 represents death and 1 represents perfect health.
  units on a scale | 0.61 (0.17)
Chronic Pain Sleep Inventory (CPSI) [Mean (Standard Deviation); unit: units on a scale] — The Chronic Pain Sleep Inventory (CPSI) is an instrument used to assess the extent to which pain interferes with sleep quality in chronic pain populations. Scores range from 0 to 100, with higher values indicating greater levels of pain-mediated sleep interference.
  units on a scale | 51.9 (30.7)
Medication Quantification Scale (MQS) III Score [Mean (Standard Deviation); unit: units on a scale] — The Medication Quantification Scale (MQS) III is used to objectively quantify and monitor pain medication use (including opioid and non-opioid medications) in chronic pain populations. The lowest possible MQS III score is 0, indicating no current usage of any analgesic drugs assessed by this instrument. It is not possible to define a maximum score value because no theoretical upper limit exists. However, higher scores reflect greater negative impacts of a pain medication regimen, and a score of 6.8 points on the MQS III is comparable to 10 daily morphine equivalents in milligrams.
  units on a scale | 6.0 (4.8)
Affected Cervical Spinal Nerve Root Levels [Count of Participants; unit: Participants]
  C4: Yes | 0
  C4: No | 33
  C5: Yes | 0
  C5: No | 33
  C6: Yes | 18
  C6: No | 15
  C7: Yes | 14
  C7: No | 19
  C8: Yes | 1
  C8: No | 32
Cervical Disc Herniation on MRI [Count of Participants; unit: Participants] — Measures whether or not a cervical disc herniation was identified on a participant's MRI prior to the procedure.
  Participants
    Yes | 11
    No | 22
Cervical Disc-Osteophyte Complex on MRI [Count of Participants; unit: Participants] — Measures whether or not a participant's MRI showed the development of osteophytes, or bone spurs, affecting their cervical disks.
  Participants
    Yes | 15
    No | 18
Cervical Foraminal Stenosis Related to Bony Elements on MRI [Count of Participants; unit: Participants] — Measures whether or not a participant's MRI showed stenosis, or narrowing, of the cervical vertebral foramen due to bone spurs.
  Participants
    Yes | 9
    No | 24
Foraminal Stenosis Severity (Park Classification) [Count of Participants; unit: Participants] — The Park classification system is as follows: Grade 0, indicating no significant stenosis or perineural fat obliteration; Grade 1 (mild), with less than 50% nerve root circumference involvement of perineural fat and no morphological change in the nerve root; Grade 2 (moderate), with greater than 50% nerve root circumference involvement of perineural fat yet without morphological change; and Grade 3 (severe), characterized by extensive perineural fat obliteration accompanied by morphological collapse of the nerve root.
  Participants
    Grade 0 or 1 | 9
    Grade 2 | 7
    Grade 3 | 17
Tobacco Use [Count of Participants; unit: Participants]
  History of tobacco use: Yes | 3
  History of tobacco use: No | 30
  Current tobacco use: Yes | 2
  Current tobacco use: No | 31
History of Depression [Count of Participants; unit: Participants]
  Yes | 9
  No | 24
History of Anxiety [Count of Participants; unit: Participants]
  Yes | 7
  No | 26

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reporting ≥50% Reduction in Index Numeric Rating Scale (NRS) Arm Pain Score
Description: Percentage of participants reporting 50% or greater improvement in index arm pain following an initial cervical transforaminal injection of steroid (CTFESI) at 1, 3, 6, and 12 months post-injection. Patient-reported arm pain intensity scores were captured at baseline and the designated follow-up time points using an 11-point Numeric Rating Scale ranging from 0 to 10, with 0 representing "no pain at all" and 10 representing "the worst pain imaginable".
Time Frame: 1 month, 3 months, 6 months, 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cervical Pain for 6 Months or Less and Scheduled for TFESI
Number analyzed (Participants) | 33
Participants
  1 month | 19
  3 months | 23
  6 months | 20
  12 months | 20

2. Secondary Outcome: Percentage of Participants Reporting ≥50% Reduction in Index Numeric Rating Scale (NRS) Neck Pain Score
Description: Percentage of participants reporting 50% or greater improvement in index neck pain following an initial cervical transforaminal injection of steroid (CTFESI) at 1, 3, 6, and 12 months post-injection. Patient-reported arm pain intensity scores were captured at baseline and the designated follow-up time points using an 11-point Numeric Rating Scale ranging from 0 to 10, with 0 representing "no pain at all" and 10 representing "the worst pain imaginable".
Time Frame: 1 month, 3 months, 6 months, 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cervical Pain for 6 Months or Less and Scheduled for TFESI
Number analyzed (Participants) | 33
Participants
  1 month | 11
  3 months | 14
  6 months | 9
  12 months | 13

3. Secondary Outcome: The Number of Participants With a ≥30% Improvement in Neck Disability Index (NDI-5)
Description: The 5-Item Neck Disability Index (NDI-5) is an assessment tool measuring patients' self-reported functional limitations due to neck pain. The range of possible scores is 0 to 24, with higher scores indicating greater functional impairment in activities of daily living.
Time Frame: 1 month, 3 months, 6 months, 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cervical Pain for 6 Months or Less and Scheduled for TFESI
Number analyzed (Participants) | 33
Participants
  1 month | 20
  3 months | 22
  6 months | 19
  12 months | 22

4. Secondary Outcome: The Number of Participants With a ≥0.03 Point Increase in EuroQol Health-Related Quality of Life (EQ-5D) Score
Description: The EuroQol Health-Related Quality of Life 5-Dimension (EQ-5D) is an instrument used in clinical and research settings to assess overall quality of life across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Scores are reported as an index ranging from 0 to 1, where 0 represents death and 1 represents perfect health.
Time Frame: 1 month, 3 months, 6 months, 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cervical Pain for 6 Months or Less and Scheduled for TFESI
Number analyzed (Participants) | 33
Participants
  1 month | 25
  3 months | 25
  6 months | 19
  12 months | 23

5. Secondary Outcome: The Number of Participants With a ≥6.8 Point Change in Medication Quantification Scale (MQS-III) Score
Description: The Medication Quantification Scale (MQS) III is used to objectively quantify and monitor pain medication use (including opioid and non-opioid medications) in chronic pain populations. The lowest possible MQS III score is 0, indicating no current usage of any analgesic drugs assessed by this instrument. It is not possible to define a maximum score value because no theoretical upper limit exists. However, higher scores reflect greater negative impacts of a pain medication regimen, and a score of 6.8 points on the MQS III is comparable to 10 daily morphine equivalents in milligrams.
Time Frame: 1 month, 3 months, 6 months, 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cervical Pain for 6 Months or Less and Scheduled for TFESI
Number analyzed (Participants) | 33
Participants
  1 month | 4
  3 months | 4
  6 months | 6
  12 months | 6

6. Secondary Outcome: The Number of Participants With a ≥30% Change in Chronic Pain Sleep Inventory (CPSI) Score
Description: The Chronic Pain Sleep Inventory (CPSI) is an instrument used to assess the extent to which pain interferes with sleep quality in chronic pain populations. Scores range from 0 to 100, with higher values indicating greater levels of pain-mediated sleep interference.
Time Frame: 1 month, 3 months, 6 months, 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cervical Pain for 6 Months or Less and Scheduled for TFESI
Number analyzed (Participants) | 33
Participants
  1 month | 9
  3 months | 12
  6 months | 5
  12 months | 7

7. Secondary Outcome: Participant Improvement in Ability to Accomplish ≥3 Key Activities From Clinical Outcome Measurement Brief Instrument (COMBI)
Description: A measure of how many participants indicated an improvement in their ability to accomplish 4 key activities: driving, exercising, sleeping and sitting.
Time Frame: 1 month, 3 months, 6 months, 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cervical Pain for 6 Months or Less and Scheduled for TFESI
Number analyzed (Participants) | 33
Participants
  1 month | 11
  3 months | 18
  6 months | 14
  12 months | 16

8. Secondary Outcome: ≥6 Patient Global Impression of Change (PGIC) Score
Description: Patient Global Impression of Change is a 7-point scale measuring participant reported satisfaction after an intervention. The outcome was measured as the percent of patients reporting a PGIC score of 6-7 (indicating "much improved" and "very much improved").
Time Frame: 1 month, 3 months, 6 months, 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cervical Pain for 6 Months or Less and Scheduled for TFESI
Number analyzed (Participants) | 33
Participants
  1 month | 18
  3 months | 21
  6 months | 15
  12 months | 18

ADVERSE EVENTS:
Time Frame: Day of procedure
Description: Any adverse events or reactions the participant experiences during and immediately after the procedure.
Arm/Group | Cervical Pain for 6 Months or Less and Scheduled for TFESI
All-Cause Mortality (participants affected / at risk) | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-13): https://cdn.clinicaltrials.gov/large-docs/83/NCT04544683/Prot_SAP_000.pdf